CLINICAL TRIAL: NCT01892319
Title: An International Non-interventional Cohort Study to Evaluate the Safety of Treatment With Levemir® (Insulin Detemir) in Pregnant Women With Diabetes Mellitus
Brief Title: An International Non-interventional Cohort Study to Evaluate the Safety of Treatment With Insulin Detemir in Pregnant Women With Diabetes Mellitus. Diabetes Pregnancy Registry
Status: Completed | Type: Observational
Sponsor: Novo Nordisk A/S (Industry)
Responsible Party: Sponsor
Other Study IDs: NN304-4016; U1111-1132-9442 (Other: WHO); ENCEPP/SDPP/4137 (Registry Identifier: EU PAS)
Record Dates: First submitted 2013-06-27; First posted 2013-07-04 (Estimated); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2 | interventions — Insulin Detemir

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All patients
  Interventions: Drug: insulin detemir; Drug: other injectable antidiabetic treatment regimens

INTERVENTIONS:
Drug: insulin detemir — Patients will be treated according to routine clinical practice at the discretion of the treating physician
Drug: other injectable antidiabetic treatment regimens — Patients will be treated according to routine clinical practice at the discretion of the treating physician

SUMMARY:
This study is conducted in Europe and Asia. The purpose of the study (Diabetes Pregnancy Registry) is to evaluate the safety of treatment with insulin detemir in pregnant women with diabetes mellitus.

ELIGIBILITY:
Inclusion Criteria: - Informed consent obtained before any data collection - Woman with a positive pregnancy test - Diabetes mellitus type 1 or 2, diagnosed prior to conception - Currently treated with Levemir® or other injectable antidiabetic treatment(s) - Unchanged basal insulin or other injectable antidiabetic treatment product (for those not treated with basal insulin) 4 weeks prior to and following conception Exclusion Criteria: - Women who have been pregnant for more than 16 weeks at baseline visit will be excluded from the study

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Women with diabetes mellitus, who are pregnant and treated with Levemir® or other injectable antidiabetic treatment regimens, and who have not changed basal insulin or other injectable antidiabetic treatment product (for those not treated with basal insulin) 4 weeks prior to and following conception will be included in the Diabetes Pregnancy Registry.
Sampling Method: Non-Probability Sample
Enrollment: 2446 (Actual)
Dates: Start 2013-09-30 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Proportion of pregnancies (Levemir® treatment), compared to pregnancies (other basal insulin treatment regimens), resulting in none of the following events: Major congenital malformations, Perinatal death, Neonatal death | Assessed up to 4 weeks after delivery

SECONDARY OUTCOMES:
Incidence of major hypoglycaemia | During pregnancy
Proportion of pregnancies complicated by pre-eclampsia | During pregnancy
Proportion of pregnancies resulting in perinatal death | Assessed 1 week after delivery
Proportion of pregnancies resulting in neonatal death | Assessed 4 weeks after delivery
Proportion of pregnancies resulting in spontaneous abortion | Assessed at pregnancy termination
Proportion of pregnancies resulting in pre-term delivery | Assessed at delivery
Height | At the age of 1 year
Weight | At the age of 1 year
Proportion with changes (progression/regression) of major congenital malformations | At the age of 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Global Clinical Registry (GCR, 1452), Study Director — Novo Nordisk A/S
Locations (80):
- Novo Nordisk Investigational Site, Zagreb, Croatia
- Finland (3):
  - Novo Nordisk Investigational Site, Pori
  - Novo Nordisk Investigational Site, Tampere
  - Novo Nordisk Investigational Site, Turku
- France (7):
  - Novo Nordisk Investigational Site, Angers
  - Novo Nordisk Investigational Site, Corbeil-Essonnes
  - Novo Nordisk Investigational Site, Lille
  - Novo Nordisk Investigational Site, Nîmes
  - Novo Nordisk Investigational Site, Paris
  - Novo Nordisk Investigational Site, Toulouse
  - Novo Nordisk Investigational Site, Valenciennes
- Germany (9):
  - Novo Nordisk Investigational Site, Bramsche
  - Novo Nordisk Investigational Site, Eisenach
  - Novo Nordisk Investigational Site, Essen
  - Novo Nordisk Investigational Site, Friedrichsthal
  - Novo Nordisk Investigational Site, Ludwigshafen
  - Novo Nordisk Investigational Site, Neuwied
  - Novo Nordisk Investigational Site, Speyer
  - Novo Nordisk Investigational Site, Stuttgart
  - Novo Nordisk Investigational Site, Sulzbach-Rosenberg
- Greece (2):
  - Novo Nordisk Investigational Site, Athens
  - Novo Nordisk Investigational Site, Nea Efkarpia - Thessaloniki
- Ireland (4):
  - Novo Nordisk Investigational Site, Castlebar
  - Novo Nordisk Investigational Site, Co. Donegal
  - Novo Nordisk Investigational Site, Dublin
  - Novo Nordisk Investigational Site, Galway
- Novo Nordisk Investigational Site, Petah Tikva, Israel
- Italy (8):
  - Novo Nordisk Investigational Site, Livorno
  - Novo Nordisk Investigational Site, Milan
  - Novo Nordisk Investigational Site, Padua
  - Novo Nordisk Investigational Site, Roma
  - Novo Nordisk Investigational Site, Sant'Andrea Delle Fratte (PG)
  - Novo Nordisk Investigational Site, Torino
  - Novo Nordisk Investigational Site, Trento
  - Novo Nordisk Investigational Site, Verona
- Malaysia (7):
  - Novo Nordisk Investigational Site, Alor Gajah
  - Novo Nordisk Investigational Site, Alor Star
  - Novo Nordisk Investigational Site, Batu Caves
  - Novo Nordisk Investigational Site, Ipoh
  - Novo Nordisk Investigational Site, Kuala Lumpur
  - Novo Nordisk Investigational Site, Putrajaya
  - Novo Nordisk Investigational Site, Seremban
- Netherlands (5):
  - Novo Nordisk Investigational Site, Amsterdam
  - Novo Nordisk Investigational Site, Apeldoorn
  - Novo Nordisk Investigational Site, Arnhem
  - Novo Nordisk Investigational Site, Eindhoven
  - Novo Nordisk Investigational Site, Utrecht
- Norway (7):
  - Novo Nordisk Investigational Site, Ålesund
  - Novo Nordisk Investigational Site, Bergen
  - Novo Nordisk Investigational Site, Gjøvik
  - Novo Nordisk Investigational Site, Hamar
  - Novo Nordisk Investigational Site, Lillehammer
  - Novo Nordisk Investigational Site, Moss
  - Novo Nordisk Investigational Site, Tønsberg
- Poland (5):
  - Novo Nordisk Investigational Site, Legnica
  - Novo Nordisk Investigational Site, Lodz
  - Novo Nordisk Investigational Site, Lubin
  - Novo Nordisk Investigational Site, Poznan
  - Novo Nordisk Investigational Site, Szczecin
- Portugal (5):
  - Novo Nordisk Investigational Site, Almada
  - Novo Nordisk Investigational Site, Amadora
  - Novo Nordisk Investigational Site, Leiria
  - Novo Nordisk Investigational Site, Lisbon
  - Novo Nordisk Investigational Site, Porto
- Romania (3):
  - Novo Nordisk Investigational Site, Timișoara, Timiș County
  - Novo Nordisk Investigational Site, Bucharest
  - Novo Nordisk Investigational Site, Galati
- Spain (5):
  - Novo Nordisk Investigational Site, Barcelona
  - Novo Nordisk Investigational Site, Madrid
  - Novo Nordisk Investigational Site, Málaga
  - Novo Nordisk Investigational Site, Seville
  - Novo Nordisk Investigational Site, Valencia
- United Kingdom (8):
  - Novo Nordisk Investigational Site, Bath
  - Novo Nordisk Investigational Site, Belfast
  - Novo Nordisk Investigational Site, Bristol
  - Novo Nordisk Investigational Site, Devon
  - Novo Nordisk Investigational Site, Glasgow
  - Novo Nordisk Investigational Site, Inverness
  - Novo Nordisk Investigational Site, Southampton
  - Novo Nordisk Investigational Site, Stevenage

REFERENCES:
- [Result] Mathiesen ER, Andersen H, Kring SI, Damm P. Design and rationale of a large, international, prospective cohort study to evaluate the occurrence of malformations and perinatal/neonatal death using insulin detemir in pregnant women with diabetes in comparison with other long-acting insulins. BMC Pregnancy Childbirth. 2017 Jan 18;17(1):38. doi: 10.1186/s12884-016-1177-4. PMID 28100192
- [Derived] Thorius IH, Petersen J, Husemoen LLN, Alibegovic AC, Gall MA, Damm P, Mathiesen ER. Glycemic Control and Risk of Congenital Malformations in Women With Type 1 Diabetes. Obstet Gynecol. 2024 Nov 1;144(5):725-732. doi: 10.1097/AOG.0000000000005722. Epub 2024 Sep 5. PMID 39236320
- [Derived] Mathiesen ER, Ali N, Alibegovic AC, Anastasiou E, Cypryk K, de Valk H, Dores J, Dunne F, Gall MA, Garcia SD, Hanaire HP, Husemoen LLN, Ivanisevic M, Kempe HP, McCance DR, Damm P. Risk of Major Congenital Malformations or Perinatal or Neonatal Death With Insulin Detemir Versus Other Basal Insulins in Pregnant Women With Preexisting Diabetes: The Real-World EVOLVE Study. Diabetes Care. 2021 Sep;44(9):2069-2077. doi: 10.2337/dc21-0472. Epub 2021 Jul 30. PMID 34330786
- See also: Clinical Trials at Novo Nordisk — http://novonordisk-trials.com